CLINICAL TRIAL: NCT02010515
Title: Clinical-Electrophysiological Risk Marker Trial Goettingen
Brief Title: An Arrhythmia Risk Predictor Trial
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Markus Zabel, Associate Professor, Head of Clinical Electrophysiology, University Medical Center Goettingen
Other Study IDs: UMG-181211
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Cardiomyopathy; Heart Failure
Keywords: sudden cardiac death; risk stratification; t-wave alternans; Holter electrocardiography; heart rate turbulence
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sinus rhythm, first ICD implantation

SUMMARY:
This prospective single-center study is an observational risk stratification trial in about 250 patients with standard indications for ICD treatment.

Implantable cardioverter defibrillators (ICD) have been shown to improve survival and current guidelines recommend their use for primary and secondary prevention of sudden cardiac death (SCD). However, a large number of patients never receive an appropriate therapy from their device. In contrast, electrical sorm and multiple ICD shocks occur in other patients.

Thus, identification of predictors for survival or ICD shocks is necessary for improved patient selection and optimized therapeutic strategies.

Risk stratification with electrocardiogram (ECG) and signal averaged ECG (SAECG), T-wave alternans (TWA) and Holter ECG including premature ventricular contractions (PVC), non-sustained VT (nsVT), heart rate variability (HRV), heart rate turbulence (HRT) and deceleration capacity, as well as clinical variables is possible, but not implemented in clinical routine in patients with ischemic or dilated cardiomyopathy and newly implanted ICD for primary or secondary prevention of SCD following current guidelines.

Patients will be prospectively followed and the predictive value of the risk markers mentioned above to predict all-cause mortality or appropriate ICD shocks will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or dilated cardiomyopathy
* sinusrhythm
* ICD indication strictly following current guidelines (primary and secondary prevention of SCD)
* Age 18 years or older

Exclusion Criteria:

* no consent
* atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic or dilated cardiomyopathy and "standard indications" for ICD treatment. "Stamdard indications" are approved and strictly follow current guidelines, the decision on ICD implantation is based on left-ventricular ejection fraction or the history of malignant arrhythmia. i.e. secondary prevention of sudden cardiac death). Implantation procedure is performed at University Medical Center Goettingen.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2008-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 2008-2013
First Appropriate ICD Shock | 2008-2013
  First ICD discharge for malignant ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, M.D., Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

REFERENCES:
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B, Blanc JJ, Budaj A, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (writing committee to develop Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Sep 5;114(10):e385-484. doi: 10.1161/CIRCULATIONAHA.106.178233. Epub 2006 Aug 25. No abstract available. PMID 16935995
- [Background] Tung R, Zimetbaum P, Josephson ME. A critical appraisal of implantable cardioverter-defibrillator therapy for the prevention of sudden cardiac death. J Am Coll Cardiol. 2008 Sep 30;52(14):1111-21. doi: 10.1016/j.jacc.2008.05.058. PMID 18804736
- [Background] Buxton AE, Lee KL, Hafley GE, Pires LA, Fisher JD, Gold MR, Josephson ME, Lehmann MH, Prystowsky EN; MUSTT Investigators. Limitations of ejection fraction for prediction of sudden death risk in patients with coronary artery disease: lessons from the MUSTT study. J Am Coll Cardiol. 2007 Sep 18;50(12):1150-7. doi: 10.1016/j.jacc.2007.04.095. Epub 2007 Sep 4. PMID 17868806
- [Background] Hohnloser SH, Ikeda T, Bloomfield DM, Dabbous OH, Cohen RJ. T-wave alternans negative coronary patients with low ejection and benefit from defibrillator implantation. Lancet. 2003 Jul 12;362(9378):125-6. doi: 10.1016/s0140-6736(03)13865-2. PMID 12867114
- [Background] Buckingham TA, Thessen CC, Stevens LL, Redd RM, Kennedy HL. Effect of conduction defects on the signal-averaged electrocardiographic determination of late potentials. Am J Cardiol. 1988 Jun 1;61(15):1265-71. doi: 10.1016/0002-9149(88)91167-8. PMID 3376884
- [Background] Bigger JT Jr, Fleiss JL, Kleiger R, Miller JP, Rolnitzky LM. The relationships among ventricular arrhythmias, left ventricular dysfunction, and mortality in the 2 years after myocardial infarction. Circulation. 1984 Feb;69(2):250-8. doi: 10.1161/01.cir.69.2.250. PMID 6690098
- [Background] Schmidt G, Malik M, Barthel P, Schneider R, Ulm K, Rolnitzky L, Camm AJ, Bigger JT Jr, Schomig A. Heart-rate turbulence after ventricular premature beats as a predictor of mortality after acute myocardial infarction. Lancet. 1999 Apr 24;353(9162):1390-6. doi: 10.1016/S0140-6736(98)08428-1. PMID 10227219
- [Background] Bauer A, Kantelhardt JW, Barthel P, Schneider R, Makikallio T, Ulm K, Hnatkova K, Schomig A, Huikuri H, Bunde A, Malik M, Schmidt G. Deceleration capacity of heart rate as a predictor of mortality after myocardial infarction: cohort study. Lancet. 2006 May 20;367(9523):1674-81. doi: 10.1016/S0140-6736(06)68735-7. PMID 16714188
- [Derived] Seegers J, Bergau L, Exposito PM, Bauer A, Fischer TH, Luthje L, Hasenfuss G, Friede T, Zabel M. Prediction of Appropriate Shocks Using 24-Hour Holter Variables and T-Wave Alternans After First Implantable Cardioverter-Defibrillator Implantation in Patients With Ischemic or Nonischemic Cardiomyopathy. Am J Cardiol. 2016 Jul 1;118(1):86-94. doi: 10.1016/j.amjcard.2016.04.016. Epub 2016 Apr 22. PMID 27189815